CLINICAL TRIAL: NCT06939673
Title: A Clinical Study of Reprise Biomedical's Miro3D Wound Matrix in the Outpatient Management of Wounds and Ulcerations
Brief Title: Study of Miro3D Wound Matrix for Healing Wounds and Ulcers in Outpatient Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reprise Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPRISE001; 20240306 (Other: WCG IRB)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcers (DFUs); Venous Leg Ulcers (VLUs); Pressure Ulcers; Surgical Wound Dehiscence (SWD); Chronic Wounds; Undermined and Tunneling Wounds
Keywords: Miro3D Wound Matrix; Acellular Wound Matrix; Porcine-Derived Scaffold; Chronic Wound Healing; Diabetic Foot Ulcer Treatment; Pressure Ulcer Management; Surgical Wound Dehiscence Therapy; Venous Leg Ulcer Treatment; Tunneling and Undermining Wounds; Complex Wound Management; Reprise Biomedical
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer; Surgical Wound Dehiscence

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive the same intervention: Miro3D Wound Matrix plus standard of care (SOC). There is no comparator or control arm. The study follows a single-arm, prospective design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Miro3D Wound Matrix plus Standard of Care (SOC) (Experimental): Participants in this single-arm study will receive Miro3D Wound Matrix in addition to standard wound care procedures. Miro3D is applied directly to the debrided wound bed. It will be applied once every 7 days for the first 4 weeks. If the wound has not closed by then, Miro3D will be applied every 14 days through week 12 or until wound closure, whichever comes first. Standard care includes debridement, dressing changes, offloading and/or compression, and infection management as needed. Weekly evaluations are performed to track healing progress.
  Interventions: Device: Acellular Porcine-Derived Wound Matrix

INTERVENTIONS:
Device: Acellular Porcine-Derived Wound Matrix — This intervention is a sterile, acellular, three-dimensional biologic scaffold derived from porcine liver tissue using a proprietary perfusion decellularization and drying process. It retains the native extracellular matrix structure and supports tissue granulation and healing in complex wounds. Miro3D is applied topically to the debrided wound bed and rehydrated prior to use. It is indicated for use in a range of chronic and complex wounds, including diabetic foot ulcers, venous leg ulcers, pressure injuries, and surgical dehiscence. In this study, it is administered in an outpatient setting alongside standard of care treatments.
  Other Names: Miro3D Wound Matrix

SUMMARY:
This clinical study is being conducted to evaluate how well the Miro3D Wound Matrix helps heal difficult wounds and ulcerations in an outpatient care setting. Miro3D is a biologic wound dressing made from porcine (pig) liver tissue. It is processed to remove all cells, creating a clean scaffold that can support the body's natural healing process. The goal of this study is to see how effective Miro3D is when used alongside standard wound care for helping wounds close and reducing pain and discomfort.

The study is designed as a post-market, proof-of-concept trial, meaning the product is already commercially available, and researchers are evaluating how it works in real-world clinical settings. A total of up to 20 adult participants will be enrolled. Participants may have wounds such as diabetic foot ulcers, venous leg ulcers, pressure ulcers, or surgical wound dehiscence. These wounds may be complex in nature, including tunneling or undermining, which often makes them more difficult to treat.

Participants will receive standard wound care along with weekly Miro3D applications for the first 4 weeks. If the wound is not fully healed after 4 weeks, Miro3D will then be applied every 2 weeks until healing is achieved or up to 12 weeks total. Throughout the study, participants will return weekly for wound assessments and to complete brief questionnaires about their pain levels and quality of life.

The main goals of the study are:

1. To measure how much the wound size shrinks (known as percent area reduction or PAR).
2. To evaluate how much healthy granulation tissue (new tissue) forms in the wound.
3. To compare healing outcomes when Miro3D is used weekly versus every two weeks.
4. To understand how the treatment affects patients' quality of life, including pain, mobility, and emotional wellbeing.

Each participant will be closely monitored by the clinical team throughout the 12-week study period. If a wound heals earlier, the participant will finish the study at that time. If the wound does not heal, the participant may return to their regular physician for follow-up care.

DETAILED DESCRIPTION:
This clinical study is a prospective, post-market, proof-of-concept trial evaluating the safety and effectiveness of Miro3D Wound Matrix, a biologically derived, acellular scaffold developed by Reprise Biomedical, in the outpatient treatment of complex wounds and ulcerations. Miro3D is made from porcine liver tissue and processed to retain a porous, three-dimensional structure that provides a supportive environment for tissue regeneration.

The study investigates Miro3D's real-world impact on wound healing in adult subjects presenting with chronic or complex wounds, including but not limited to diabetic foot ulcers (DFUs), pressure ulcers, venous leg ulcers (VLUs), and surgical wound dehiscence (SWD). These types of wounds are often difficult to treat, particularly when they exhibit features like tunneling or undermining. The matrix is applied in conjunction with standard of care (SOC) therapies such as cleansing, offloading, compression, debridement, and the use of secondary dressings.

Up to 20 adult participants will be enrolled at outpatient clinical sites under the supervision of a principal investigator. The study includes both a screening phase and a 12-week treatment phase. There is no run-in or washout period. Eligible subjects are identified based on criteria including wound size (1-40 cm²), duration, location, vascular perfusion, and willingness to adhere to follow-up and offloading instructions. Subjects with third-degree burns, active untreated osteomyelitis, malignancy, or known porcine allergy, among other conditions, are excluded.

Each subject will receive Miro3D applied weekly for the first four weeks. If healing has not occurred at that point, Miro3D is reapplied every two weeks for up to twelve weeks or until the wound is fully closed. Wound healing is assessed weekly through manual measurements, photographs, and depth probing. The primary study endpoint is percentage area reduction (PAR) and granulation tissue formation at 4 and 12 weeks.

Secondary endpoints include changes from baseline in patient-reported quality of life (QOL) using the Wound-QOL questionnaire, and pain intensity assessed using a visual analog scale (VAS). These questionnaires are completed weekly to gauge the impact of treatment on physical function, emotional wellbeing, pain, odor, and social engagement. In the event of premature withdrawal, efforts are made to gather final QOL and pain assessments.

Subjects attend weekly study visits and may be seen for additional unscheduled visits at the investigator's discretion (e.g., for dressing changes). If the wound heals before 12 weeks, the subject exits the study. If the wound remains open, the subject exits after the final assessment and may return to their standard treating provider.

The study also closely monitors adverse events (AEs), serious adverse events (SAEs), and unanticipated adverse device effects (UADEs). Investigators assess each event's relationship to the study product and report them to the sponsor and IRB as required. All safety data are collected throughout the study and monitored by the study team and sponsor.

The data collected include subject demographics, medical and surgical history, wound type and size, infection status, tissue characteristics, exudate volume, and treatment regimen. These data are documented in source documents and transcribed into study-specific Case Report Forms (CRFs). Statistical analysis will be performed using summary statistics to evaluate wound closure rates, healing trajectories, and possible correlations between treatment schedule and healing outcomes.

As a post-market study, this trial does not require an Investigational Device Exemption (IDE) and is conducted in compliance with Good Clinical Practice (GCP), the Health Insurance Portability and Accountability Act (HIPAA), and FDA guidelines. It has been approved by an Institutional Review Board (IRB), and informed consent is required from all participants prior to enrollment.

By evaluating Miro3D in real-world outpatient conditions, this study aims to provide evidence on its ability to promote healing in challenging wounds. The findings may help guide future treatment approaches and inform larger clinical trials focused on specific wound types.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older and able to provide informed consent.
2. Has an open wound or ulceration, preferably with tunneling or undermining.
3. If multiple wounds/ulcerations are present, only one will be selected for Miro3D treatment.
4. Other wounds must be ≥2 cm away from the study wound.
5. Wound should be debrided with a clinical goal of healing, even if some infection remains.
6. Previous infections must be adequately treated and controlled (per IDSA guidelines).
7. Willing and able to comply with offloading and/or compression requirements.
8. Must have a stable living environment for wound care adherence.
9. Study wound must have a clean base free of devitalized tissue or debris at the time of Miro3D placement.
10. Provides consent for digital photo documentation.

Exclusion Criteria:

1. Active, untreated osteomyelitis.
2. Malignancy or vasculitis at the wound site.
3. Undergoing chemotherapy.
4. On dialysis.
5. Use of investigational drugs or therapies within 30 days before screening.
6. Conditions that significantly impair study adherence or known history of medical non-compliance.
7. Known sensitivity to porcine materials.
8. Third-degree burns.
9. Worsening ischemia or gangrene at screening.
10. Prior radiation to the study wound site.
11. Exposed hardware, implants, or fixation devices in the study wound.
12. Receiving palliative or comfort care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Area Reduction (PAR) and Granulation Tissue Formation at 4 and 12 Weeks | 4 weeks and 12 weeks post-initial treatment
  The primary outcome is the measurement of the wound or ulcer's percent area reduction (PAR) and granulation tissue formation at week 4 and week 12. This is used to evaluate healing progression and the effectiveness of Miro3D. Measurements are taken using a ruler for length and width, and a probe for depth. Granulation is assessed visually by the clinical team.

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) Using Wound-QOL Instrument | Baseline and weekly through 12 weeks or until wound closure
  Subject-reported QOL will be assessed at each visit using the Wound-QOL questionnaire. This tool evaluates the impact of the wound on domains such as pain, odor, physical functioning, mobility, emotional wellbeing, and social isolation.
Change in Pain Levels Using Visual Analog Scale (VAS) | Baseline and weekly through 12 weeks or until wound closure
  Pain intensity is assessed weekly using a 0-10 VAS, where 0 represents no pain and 10 represents the worst possible pain.

OTHER OUTCOMES:
Safety and Tolerability: Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Device Effects (UADEs) | From informed consent through 30 days after final study visit
  The frequency and severity of adverse events, including product-related effects such as inflammation, irritation, or infection, will be recorded. Events will be assessed for seriousness, expectedness, and relatedness to the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Snyder, DPM, Principal Investigator — Barry University
Locations (2):
- United States (2):
  - West Boca Center for Wound Healing, Coconut Creek, Florida
  - Barry University Clinical Research, Tamarac, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith ME, Totten A, Hickam DH, Fu R, Wasson N, Rahman B, Motu'apuaka M, Saha S. Pressure ulcer treatment strategies: a systematic comparative effectiveness review. Ann Intern Med. 2013 Jul 2;159(1):39-50. doi: 10.7326/0003-4819-159-1-201307020-00007. PMID 23817703
- [Background] Raghav A, Khan ZA, Labala RK, Ahmad J, Noor S, Mishra BK. Financial burden of diabetic foot ulcers to world: a progressive topic to discuss always. Ther Adv Endocrinol Metab. 2018 Jan;9(1):29-31. doi: 10.1177/2042018817744513. Epub 2017 Dec 12. PMID 29344337
- [Background] Padula WV, Delarmente BA. The national cost of hospital-acquired pressure injuries in the United States. Int Wound J. 2019 Jun;16(3):634-640. doi: 10.1111/iwj.13071. Epub 2019 Jan 28. PMID 30693644
- [Background] Mervis JS, Phillips TJ. Pressure ulcers: Pathophysiology, epidemiology, risk factors, and presentation. J Am Acad Dermatol. 2019 Oct;81(4):881-890. doi: 10.1016/j.jaad.2018.12.069. Epub 2019 Jan 18. PMID 30664905
- [Background] Kruger EA, Pires M, Ngann Y, Sterling M, Rubayi S. Comprehensive management of pressure ulcers in spinal cord injury: current concepts and future trends. J Spinal Cord Med. 2013 Nov;36(6):572-85. doi: 10.1179/2045772313Y.0000000093. Epub 2013 May 21. PMID 24090179
- [Background] Geriatric Medicine Gerontology Chapter 30 - Pressure Ulcers. (n.d.). Retrieved from Johns Hopkins: https://www.hopkinsmedicine.org/geriatric_medicine_gerontology/_downloads/readings/section8.pdf
- [Background] Bauer K, Rock K, Nazzal M, Jones O, Qu W. Pressure Ulcers in the United States' Inpatient Population From 2008 to 2012: Results of a Retrospective Nationwide Study. Ostomy Wound Manage. 2016 Nov;62(11):30-38. PMID 27861135
- See also: Miro3D Wound Matrix product webpage — https://reprisebio.com/miro3d/